CLINICAL TRIAL: NCT06112951
Title: The Use of Extracorporeal Photopheresis as Immunomodulatory Therapy of Subclinical Antibody-mediated Rejection After Lung Transplantation: a Prospective RCT
Brief Title: A Prospective Randomized Trial of ECP in Subclinical AMR
Acronym: EUROEXPORT-DSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alberto Benazzo, Priv. Doz. Dr. Alberto Benazzo, PhD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1578/2023
Record Dates: First submitted 2023-10-09; First posted 2023-11-02 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Antibody-mediated Rejection; Lung Transplant Rejection
MeSH Terms: interventions — Photopheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Treatment group will receive extracorporeal photopheresis. First, a two-day treatment cycle will be performed once every second week for the first two months. Then, a two-day treatment cycle will be performed once a month for 6 months.
  Interventions: Procedure: Extracorporeal Photopheresis
- Control Group (No Intervention): Control group will be observed and no active treatment will be administered. This is our standard of care in the studied clinical situation.

INTERVENTIONS:
Procedure: Extracorporeal Photopheresis — Patients randomized into the interventional group will receive ECP. ECP will be started within one week after randomization. Initially a two-day treatment cycle will be performed once every second week for the first two months. Then, a two-day treatment cycle will be performed once a month for 6 months.
  Arms: Treatment Group

SUMMARY:
The goal of this clinical trial is to evaluate the therapeutic effect of extracorporeal photopheresis in subclinical antibody-mediated rejection after lung transplantation.The main questions it aims to answer are:

1. Does ECP therapy result in a significant reduction in MFI (Mean Fluorescence Intensity) from the baseline MFI in clinically stable patients with persistent (>6 months) dnDSAs (MFI>1000)?
2. What is the impact of ECP therapy on the following outcomes in these patients: ACR, clinical AMR, CLAD, infections, drop-out rate, survival, adverse events?

Participants will be randomized into two groups. Each group will include 40 patients. The control group will be observed and no active treatment will be administered. The treatment group will receive extracorporeal photopheresis. First, a two-day treatment cycle will be performed once every second week for the first two months. Then, a two-day treatment cycle will be performed once a month for 6 months.

Researchers will compare the two groups regarding: MFI value, development of ACR, clinical AMR, CLAD, infections, survival, adverse events, immunophenotyping, miRNA expression profiling, cytokine expression, gene expression signature of PBMCs and proteomic characterization.

DETAILED DESCRIPTION:
Donor-specific antibodies (DSA) and antibody-mediated rejection have gained significant attention recently due to their serious consequences, but there are limited effective treatments for persistent DSAs in patients without graft dysfunction due to their associated severe side effects. Our center demonstrated that extracorporeal photopheresis (ECP) can potentially reduce the mean fluorescence intensity of dnDSAs in recipients with antibody-mediated rejection (AMR), suggesting it as a safe option for treating subclinical AMR with dnDSAs and inducing tolerogenic immunomodulation in this complex population.

The hypothesis underlying the proposed randomized controlled trial is that ECP might have the potential to reduce the burden of de novo donor-specific antibodies after lung transplantation, by modulating host humoral alloresponse and promoting tolerance, without provoking side effects.

Our primary objective is to evaluate the therapeutic effect of ECP in terms of reduction of dnDSAs titer in clinically stable patients with persistent (>6 months) dnDSAs (MFI>1000). As secondary objective, we intend to assess the therapeutic effect of ECP on incidence of clinical AMR, ACR, CLAD, survival and occurrence of infectious complications as well as the rate of adverse effects. Our experimental objectives are to provide an in-depth analysis of the immunological effects of ECP.

80 patients with persistent dnDSAs (> 3 months) with a MFI > 1000 will be randomized into two groups. Each group will include 40 patients. Patients will be stratified according to the presence of HLA-DQ. The control group will be observed and no active treatment will be administered. This is our standard of care in the studied clinical situation. Treatment group will receive extracorporeal photopheresis. First, a two-day treatment cycle will be performed once every second week for the first two months. Then, a two-day treatment cycle will be performed once a month for 6 months. To elucidate the specific mechanisms of ECP in modulating humoral alloresponse, a series of studies are planned: 1) flow cytometric immunophenotyping, 2) miRNA expression profiling, 3) cytokine expression, 4) gene expression signature of PBMCs, 5) proteomic characterization.

The proposed study aims to address this clinical need by investigating the effects of a safe therapeutic modality such as ECP. This study may have a dual benefit: first, it may reduce the burden of dnDSAs in lung transplant recipients, thereby reducing the incidence of antibody-mediated rejection, and second, it may promote host tolerance to the graft. In addition, we will investigate the immunomodulatory mechanisms of ECP in the context of humoral allogeneic response, which has not been previously investigated.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral lung transplantation
* dnDSAs > 3 months with a MFI > 1000
* No signs of allograft dysfunction
* Alemtuzumab induction therapy

Exclusion Criteria:

* Inclusion in other studies
* Retransplantation
* Multi-organ transplantation
* > 12 months after transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of dnDSA titer from baseline MFI | 6 months
  Difference of MFI values at the start and at the end of the six month period

SECONDARY OUTCOMES:
Incidence of clinical AMR, ACR, CLAD, survival, infectious complications, adverse effects | 6 months
  Incidence of clinical AMR, ACR, CLAD, survival, infectious complications, adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Benazzo, MD PhD, Principal Investigator — Medical University of Vienna
Locations (7):
- Medical University of Vienna, Vienna, Austria
- UZ Leuven, Leuven, Belgium
- University Hospital Center Zagreb, Zagreb, Croatia
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark
- Hôpital Foch, Suresnes, France
- Policlinico San Matteo Pavia Fondazione IRCCS, Pavia, Italy
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Chambers DC, Perch M, Zuckermann A, Cherikh WS, Harhay MO, Hayes D Jr, Hsich E, Khush KK, Potena L, Sadavarte A, Lindblad K, Singh TP, Stehlik J; International Society for Heart and Lung Transplantation. The International Thoracic Organ Transplant Registry of the International Society for Heart and Lung Transplantation: Thirty-eighth adult lung transplantation report - 2021; Focus on recipient characteristics. J Heart Lung Transplant. 2021 Oct;40(10):1060-1072. doi: 10.1016/j.healun.2021.07.021. Epub 2021 Jul 31. PMID 34446355
- [Background] Benazzo A, Auner S, Boehm PM, Morscher A, Schwarz S, Vidmar B, Dzubur F, Schweiger T, Hoda AM, Moser B, Matilla JR, Murakozy G, Lang G, Taghavi S, Klepetko W, Hoetzenecker K, Jaksch P. Outcomes with alemtuzumab induction therapy in lung transplantation: a comprehensive large-scale single-center analysis. Transpl Int. 2021 Dec;34(12):2633-2643. doi: 10.1111/tri.14153. Epub 2021 Nov 16. PMID 34738249
- [Background] Iasella CJ, Ensor CR, Marrari M, Mangiola M, Xu Q, Nolley E, Moore CA, Morrell MR, Pilewski JM, Sanchez PG, McDyer JF, Zeevi A. Donor-specific antibody characteristics, including persistence and complement-binding capacity, increase risk for chronic lung allograft dysfunction. J Heart Lung Transplant. 2020 Dec;39(12):1417-1425. doi: 10.1016/j.healun.2020.09.003. Epub 2020 Sep 10. PMID 32981841
- [Background] Benazzo A, Worel N, Schwarz S, Just U, Nechay A, Lambers C, Bohmig G, Fischer G, Koren D, Murakozy G, Knobler R, Klepetko W, Hoetzenecker K, Jaksch P. Outcome of Extracorporeal Photopheresis as an Add-On Therapy for Antibody-Mediated Rejection in Lung Transplant Recipients. Transfus Med Hemother. 2020 Jun;47(3):205-213. doi: 10.1159/000508170. Epub 2020 May 5. PMID 32595425
- [Background] Gasparro FP, Felli A, Schmitt IM. Psoralen photobiology: the relationship between DNA damage, chromatin structure, transcription, and immunogenic effects. Recent Results Cancer Res. 1997;143:101-27. doi: 10.1007/978-3-642-60393-8_8. No abstract available. PMID 8912415
- [Background] Kurts C, Kosaka H, Carbone FR, Miller JF, Heath WR. Class I-restricted cross-presentation of exogenous self-antigens leads to deletion of autoreactive CD8(+) T cells. J Exp Med. 1997 Jul 21;186(2):239-45. doi: 10.1084/jem.186.2.239. PMID 9221753
- [Background] Maeda A, Schwarz A, Bullinger A, Morita A, Peritt D, Schwarz T. Experimental extracorporeal photopheresis inhibits the sensitization and effector phases of contact hypersensitivity via two mechanisms: generation of IL-10 and induction of regulatory T cells. J Immunol. 2008 Nov 1;181(9):5956-62. doi: 10.4049/jimmunol.181.9.5956. PMID 18941184
- [Background] Maeda A, Schwarz A, Kernebeck K, Gross N, Aragane Y, Peritt D, Schwarz T. Intravenous infusion of syngeneic apoptotic cells by photopheresis induces antigen-specific regulatory T cells. J Immunol. 2005 May 15;174(10):5968-76. doi: 10.4049/jimmunol.174.10.5968. PMID 15879089
- [Background] Edelson RL. Mechanistic insights into extracorporeal photochemotherapy: efficient induction of monocyte-to-dendritic cell maturation. Transfus Apher Sci. 2014 Jun;50(3):322-9. doi: 10.1016/j.transci.2013.07.031. Epub 2013 Aug 8. PMID 23978554
- [Background] Knobler R. Extracorporeal photochemotherapy--present and future. Vox Sang. 2000;78 Suppl 2:197-201. PMID 10938952
- [Background] Teruel Montoya R, López-Godino O, Garcia-Barbera N, et al. Identification of Circulating microRNA Signatures As Potential Noninvasive Biomarkers for Prediction to Response to Extracorporeal Photoapheresis in Patients with Graft Versus Host Disease. Blood 2019;134:4466-.
- [Background] Bozzini S, Del Fante C, Morosini M, Berezhinskiy HO, Auner S, Cattaneo E, Della Zoppa M, Pandolfi L, Cacciatore R, Perotti C, Hoetzenecker K, Jaksch P, Benazzo A, Meloni F. Mechanisms of Action of Extracorporeal Photopheresis in the Control of Bronchiolitis Obliterans Syndrome (BOS): Involvement of Circulating miRNAs. Cells. 2022 Mar 25;11(7):1117. doi: 10.3390/cells11071117. PMID 35406680
- [Background] Morrell MR, Despotis GJ, Lublin DM, Patterson GA, Trulock EP, Hachem RR. The efficacy of photopheresis for bronchiolitis obliterans syndrome after lung transplantation. J Heart Lung Transplant. 2010 Apr;29(4):424-31. doi: 10.1016/j.healun.2009.08.029. Epub 2009 Oct 22. PMID 19853479
- [Background] Jaksch P, Scheed A, Keplinger M, Ernst MB, Dani T, Just U, Nahavandi H, Klepetko W, Knobler R. A prospective interventional study on the use of extracorporeal photopheresis in patients with bronchiolitis obliterans syndrome after lung transplantation. J Heart Lung Transplant. 2012 Sep;31(9):950-7. doi: 10.1016/j.healun.2012.05.002. PMID 22884382
- [Background] Greer M, Liu B, Magnusson JM, Fuehner T, Schmidt BMW, Deluca D, Falk C, Ius F, Welte T. Assessing treatment outcomes in CLAD: The Hannover-extracorporeal photopheresis model. J Heart Lung Transplant. 2023 Feb;42(2):209-217. doi: 10.1016/j.healun.2022.09.022. Epub 2022 Oct 5. PMID 37071121
- [Background] Rose EA, Barr ML, Xu H, Pepino P, Murphy MP, McGovern MA, Ratner AJ, Watkins JF, Marboe CC, Berger CL. Photochemotherapy in human heart transplant recipients at high risk for fatal rejection. J Heart Lung Transplant. 1992 Jul-Aug;11(4 Pt 1):746-50. PMID 1498142
- [Background] Barr ML, Baker CJ, Schenkel FA, McLaughlin SN, Stouch BC, Starnes VA, Rose EA. Prophylactic photopheresis and chronic rejection: effects on graft intimal hyperplasia in cardiac transplantation. Clin Transplant. 2000 Apr;14(2):162-6. doi: 10.1034/j.1399-0012.2000.140211.x. PMID 10770423
- [Background] Hidalgo LG, Campbell PM, Sis B, Einecke G, Mengel M, Chang J, Sellares J, Reeve J, Halloran PF. De novo donor-specific antibody at the time of kidney transplant biopsy associates with microvascular pathology and late graft failure. Am J Transplant. 2009 Nov;9(11):2532-41. doi: 10.1111/j.1600-6143.2009.02800.x. PMID 19843031
- [Background] Zeevi A, Lunz J, Feingold B, Shullo M, Bermudez C, Teuteberg J, Webber S. Persistent strong anti-HLA antibody at high titer is complement binding and associated with increased risk of antibody-mediated rejection in heart transplant recipients. J Heart Lung Transplant. 2013 Jan;32(1):98-105. doi: 10.1016/j.healun.2012.09.021. Epub 2012 Nov 9. PMID 23142561
- [Background] Safavi S, Robinson DR, Soresi S, Carby M, Smith JD. De novo donor HLA-specific antibodies predict development of bronchiolitis obliterans syndrome after lung transplantation. J Heart Lung Transplant. 2014 Dec;33(12):1273-81. doi: 10.1016/j.healun.2014.07.012. Epub 2014 Jul 21. PMID 25130554
- [Background] Girnita AL, Duquesnoy R, Yousem SA, Iacono AT, Corcoran TE, Buzoianu M, Johnson B, Spichty KJ, Dauber JH, Burckart G, Griffith BP, McCurry KR, Zeevi A. HLA-specific antibodies are risk factors for lymphocytic bronchiolitis and chronic lung allograft dysfunction. Am J Transplant. 2005 Jan;5(1):131-8. doi: 10.1111/j.1600-6143.2004.00650.x. PMID 15636621
- [Background] Sundaresan S, Mohanakumar T, Smith MA, Trulock EP, Lynch J, Phelan D, Cooper JD, Patterson GA. HLA-A locus mismatches and development of antibodies to HLA after lung transplantation correlate with the development of bronchiolitis obliterans syndrome. Transplantation. 1998 Mar 15;65(5):648-53. doi: 10.1097/00007890-199803150-00008. PMID 9521198
- [Background] Morrell MR, Patterson GA, Trulock EP, Hachem RR. Acute antibody-mediated rejection after lung transplantation. J Heart Lung Transplant. 2009 Jan;28(1):96-100. doi: 10.1016/j.healun.2008.09.013. Epub 2008 Dec 4. PMID 19134538
- [Background] Roux A, Thomas KA, Sage E, Suberbielle-Boissel C, Beaumont-Azuar L, Parquin F, Le Guen M, Harre N, Hamid AM, Reed EF. Donor-specific HLA antibody-mediated complement activation is a significant indicator of antibody-mediated rejection and poor long-term graft outcome during lung transplantation: a single center cohort study. Transpl Int. 2018 Jul;31(7):761-772. doi: 10.1111/tri.13149. Epub 2018 Apr 22. PMID 29537702
- [Background] Hachem RR, Tiriveedhi V, Patterson GA, Aloush A, Trulock EP, Mohanakumar T. Antibodies to K-alpha 1 tubulin and collagen V are associated with chronic rejection after lung transplantation. Am J Transplant. 2012 Aug;12(8):2164-71. doi: 10.1111/j.1600-6143.2012.04079.x. Epub 2012 May 8. PMID 22568593
- [Background] Witt CA, Gaut JP, Yusen RD, Byers DE, Iuppa JA, Bennett Bain K, Alexander Patterson G, Mohanakumar T, Trulock EP, Hachem RR. Acute antibody-mediated rejection after lung transplantation. J Heart Lung Transplant. 2013 Oct;32(10):1034-40. doi: 10.1016/j.healun.2013.07.004. Epub 2013 Aug 13. PMID 23953920
- [Background] Tinckam KJ, Keshavjee S, Chaparro C, Barth D, Azad S, Binnie M, Chow CW, de Perrot M, Pierre AF, Waddell TK, Yasufuku K, Cypel M, Singer LG. Survival in sensitized lung transplant recipients with perioperative desensitization. Am J Transplant. 2015 Feb;15(2):417-26. doi: 10.1111/ajt.13076. PMID 25612494
- [Background] Hachem RR, Yusen RD, Meyers BF, Aloush AA, Mohanakumar T, Patterson GA, Trulock EP. Anti-human leukocyte antigen antibodies and preemptive antibody-directed therapy after lung transplantation. J Heart Lung Transplant. 2010 Sep;29(9):973-80. doi: 10.1016/j.healun.2010.05.006. Epub 2010 Jun 16. PMID 20558084
- [Background] Keller M, Yang S, Ponor L, Bon A, Cochrane A, Philogene M, Bush E, Shah P, Mathew J, Brown AW, Kong H, Charya A, Luikart H, Nathan SD, Khush KK, Jang M, Agbor-Enoh S. Preemptive treatment of de novo donor-specific antibodies in lung transplant patients reduces subsequent risk of chronic lung allograft dysfunction or death. Am J Transplant. 2023 Apr;23(4):559-564. doi: 10.1016/j.ajt.2022.12.019. Epub 2023 Jan 19. PMID 36732088
- [Background] Loupy A, Lefaucheur C. Antibody-Mediated Rejection of Solid-Organ Allografts. N Engl J Med. 2018 Sep 20;379(12):1150-1160. doi: 10.1056/NEJMra1802677. No abstract available. PMID 30231232
- [Background] Levine DJ, Glanville AR, Aboyoun C, Belperio J, Benden C, Berry GJ, Hachem R, Hayes D Jr, Neil D, Reinsmoen NL, Snyder LD, Sweet S, Tyan D, Verleden G, Westall G, Yusen RD, Zamora M, Zeevi A. Antibody-mediated rejection of the lung: A consensus report of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2016 Apr;35(4):397-406. doi: 10.1016/j.healun.2016.01.1223. Epub 2016 Feb 10. PMID 27044531
- [Background] Wang L, Ni M, Huckelhoven-Krauss A, Sellner L, Hoffmann JM, Neuber B, Luft T, Hegenbart U, Schonland S, Kleist C, Sill M, Chen BA, Wuchter P, Eckstein V, Kruger W, Hilgendorf I, Yerushalmi R, Nagler A, Muller-Tidow C, Ho AD, Dreger P, Schmitt M, Schmitt A. Modulation of B Cells and Homing Marker on NK Cells Through Extracorporeal Photopheresis in Patients With Steroid-Refractory/Resistant Graft-Vs.-Host Disease Without Hampering Anti-viral/Anti-leukemic Effects. Front Immunol. 2018 Oct 8;9:2207. doi: 10.3389/fimmu.2018.02207. eCollection 2018. PMID 30349527
- [Background] Bladon J, Taylor P. Extracorporeal photopheresis reduces the number of mononuclear cells that produce pro-inflammatory cytokines, when tested ex-vivo. J Clin Apher. 2002;17(4):177-82. doi: 10.1002/jca.10039. PMID 12494410
- [Background] Li W, Gauthier JM, Higashikubo R, Hsiao HM, Tanaka S, Vuong L, Ritter JH, Tong AY, Wong BW, Hachem RR, Puri V, Bharat A, Krupnick AS, Hsieh CS, Baldwin WM 3rd, Kelly FL, Palmer SM, Gelman AE, Kreisel D. Bronchus-associated lymphoid tissue-resident Foxp3+ T lymphocytes prevent antibody-mediated lung rejection. J Clin Invest. 2019 Feb 1;129(2):556-568. doi: 10.1172/JCI122083. Epub 2018 Dec 18. PMID 30561386
- [Background] Luo Y, Luo F, Zhang K, Wang S, Zhang H, Yang X, Shang W, Wang J, Wang Z, Pang X, Feng Y, Liu L, Xie H, Feng G, Li J. Elevated Circulating IL-10 Producing Breg, but Not Regulatory B Cell Levels, Restrain Antibody-Mediated Rejection After Kidney Transplantation. Front Immunol. 2021 Jan 28;11:627496. doi: 10.3389/fimmu.2020.627496. eCollection 2020. PMID 33584730
- [Background] Budde H, Berntsch U, Riggert J, Legler TJ. In vitro effects of different 8-methoxypsoralen treatment protocols for extracorporeal photopheresis on mononuclear cells. Cent Eur J Immunol. 2017;42(1):1-9. doi: 10.5114/ceji.2017.67312. Epub 2017 May 8. PMID 28680325
- [Background] Baskaran G, Tiriveedhi V, Ramachandran S, Aloush A, Grossman B, Hachem R, Mohanakumar T. Efficacy of extracorporeal photopheresis in clearance of antibodies to donor-specific and lung-specific antigens in lung transplant recipients. J Heart Lung Transplant. 2014 Sep;33(9):950-6. doi: 10.1016/j.healun.2014.04.020. Epub 2014 May 9. PMID 24906794
- [Background] McKinnon KM. Flow Cytometry: An Overview. Curr Protoc Immunol. 2018 Feb 21;120:5.1.1-5.1.11. doi: 10.1002/cpim.40. PMID 29512141
- [Background] Pitoiset F, Barbie M, Monneret G, Braudeau C, Pochard P, Pellegrin I, Trauet J, Labalette M, Klatzmann D, Rosenzwajg M. A standardized flow cytometry procedure for the monitoring of regulatory T cells in clinical trials. Cytometry B Clin Cytom. 2018 Sep;94(5):621-626. doi: 10.1002/cyto.b.21622. Epub 2018 Jan 23. PMID 29316248
- [Background] Correia RP, Rajab A, Bento LC, Alexandre AM, Vaz AC, Schimidell D, Pedro EC, Perin FS, Nozawa ST, Barroso RS, Bacal NS. A ten-color tube with dried antibody reagents for the screening of hematological malignancies. Int J Lab Hematol. 2018 Apr;40(2):136-143. doi: 10.1111/ijlh.12753. Epub 2017 Oct 4. PMID 28980400
- [Background] Rajab A, Axler O, Leung J, Wozniak M, Porwit A. Ten-color 15-antibody flow cytometry panel for immunophenotyping of lymphocyte population. Int J Lab Hematol. 2017 May;39 Suppl 1:76-85. doi: 10.1111/ijlh.12678. PMID 28447425
- [Background] Ensor CR, Yousem SA, Marrari M, Morrell MR, Mangiola M, Pilewski JM, D'Cunha J, Wisniewski SR, Venkataramanan R, Zeevi A, McDyer JF. Proteasome Inhibitor Carfilzomib-Based Therapy for Antibody-Mediated Rejection of the Pulmonary Allograft: Use and Short-Term Findings. Am J Transplant. 2017 May;17(5):1380-1388. doi: 10.1111/ajt.14222. Epub 2017 Mar 9. PMID 28173620
- [Background] Verleden GM, Glanville AR, Lease ED, Fisher AJ, Calabrese F, Corris PA, Ensor CR, Gottlieb J, Hachem RR, Lama V, Martinu T, Neil DAH, Singer LG, Snell G, Vos R. Chronic lung allograft dysfunction: Definition, diagnostic criteria, and approaches to treatment-A consensus report from the Pulmonary Council of the ISHLT. J Heart Lung Transplant. 2019 May;38(5):493-503. doi: 10.1016/j.healun.2019.03.009. Epub 2019 Apr 3. No abstract available. PMID 30962148
- [Background] Glanville AR, Verleden GM, Todd JL, Benden C, Calabrese F, Gottlieb J, Hachem RR, Levine D, Meloni F, Palmer SM, Roman A, Sato M, Singer LG, Tokman S, Verleden SE, von der Thusen J, Vos R, Snell G. Chronic lung allograft dysfunction: Definition and update of restrictive allograft syndrome-A consensus report from the Pulmonary Council of the ISHLT. J Heart Lung Transplant. 2019 May;38(5):483-492. doi: 10.1016/j.healun.2019.03.008. Epub 2019 Apr 3. No abstract available. PMID 31027539
- [Background] Stewart S, Fishbein MC, Snell GI, Berry GJ, Boehler A, Burke MM, Glanville A, Gould FK, Magro C, Marboe CC, McNeil KD, Reed EF, Reinsmoen NL, Scott JP, Studer SM, Tazelaar HD, Wallwork JL, Westall G, Zamora MR, Zeevi A, Yousem SA. Revision of the 1996 working formulation for the standardization of nomenclature in the diagnosis of lung rejection. J Heart Lung Transplant. 2007 Dec;26(12):1229-42. doi: 10.1016/j.healun.2007.10.017. PMID 18096473
- [Background] Berry G, Burke M, Andersen C, Angelini A, Bruneval P, Calabrese F, Fishbein MC, Goddard M, Leone O, Maleszewski J, Marboe C, Miller D, Neil D, Padera R, Rassl D, Revello M, Rice A, Stewart S, Yousem SA. Pathology of pulmonary antibody-mediated rejection: 2012 update from the Pathology Council of the ISHLT. J Heart Lung Transplant. 2013 Jan;32(1):14-21. doi: 10.1016/j.healun.2012.11.005. No abstract available. PMID 23260701
- [Background] Marques MB, Tuncer HH. Photopheresis in solid organ transplant rejection. J Clin Apher. 2006 Apr;21(1):72-7. doi: 10.1002/jca.20089. PMID 16619230
- [Background] Benazzo A, Bozzini S, Auner S, Berezhinskiy HO, Watzenboeck ML, Schwarz S, Schweiger T, Klepetko W, Wekerle T, Hoetzenecker K, Meloni F, Jaksch P. Differential expression of circulating miRNAs after alemtuzumab induction therapy in lung transplantation. Sci Rep. 2022 Apr 30;12(1):7072. doi: 10.1038/s41598-022-10866-w. PMID 35490174
- [Background] Benazzo A, Cho A, Nechay A, Schwarz S, Frommlet F, Wekerle T, Hoetzenecker K, Jaksch P. Combined low-dose everolimus and low-dose tacrolimus after Alemtuzumab induction therapy: a randomized prospective trial in lung transplantation. Trials. 2021 Jan 4;22(1):6. doi: 10.1186/s13063-020-04843-9. PMID 33397442
- [Background] Meier F, Brunner AD, Frank M, Ha A, Bludau I, Voytik E, Kaspar-Schoenefeld S, Lubeck M, Raether O, Bache N, Aebersold R, Collins BC, Rost HL, Mann M. diaPASEF: parallel accumulation-serial fragmentation combined with data-independent acquisition. Nat Methods. 2020 Dec;17(12):1229-1236. doi: 10.1038/s41592-020-00998-0. Epub 2020 Nov 30. PMID 33257825
- [Background] Grogan KE. How the entire scientific community can confront gender bias in the workplace. Nat Ecol Evol. 2019 Jan;3(1):3-6. doi: 10.1038/s41559-018-0747-4. No abstract available. PMID 30478306